CLINICAL TRIAL: NCT07347197
Title: A Phase I/II Study of Endocardial Delivery for Myocardial Regeneration Using Human Induced Pluripotent Stem (iPS) Cell-derived Cardiomyocyte Spheroids for Heart Failure Reduced Ejection Fraction
Brief Title: Endocardial Delivery for Myocardial Regeneration Using Allogeneic iPSC-derived Cardiomyocyte Spheroids for HF With Systolic Dysfunction (EMERALD Study)
Acronym: EMERALD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heartseed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-005-01
Record Dates: First submitted 2025-12-27; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Ischemic Heart Failure; Ischemic Heart Disease; Dilated Cardiomyopathy (DCM)
Keywords: Heart Failure; Ischemic heart failure; Ischemic Heart Disease; Dilated Cardiomyopathy (DCM); iPSC; cell therapy
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): HS-005 administration
  Interventions: Combination Product: HS-005

INTERVENTIONS:
Combination Product: HS-005 — Human (allogeneic) iPS-cell-derived cardiomyocyte spheroids (HS-001CS) transplantation with endocardial delivery systems

SUMMARY:
The purpose of this clinical study is to evaluate the safety and efficacy of endocardial delivery of HS-001 CS into severe heart failure patients with reduced ejection fraction for 26 weeks after transplantation.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase I/II study in 14 severe heart failure patients with reduced ejection fraction.

After screening period is completed, subjects undergo HS-001 CS transplantation by endocardial delivery. After transplantation, subjects take immunosuppressant and have efficacy/safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resting left ventricular ejection fraction (LVEF) ≦40% based on institutional assessment on screening echocardiographic assessment
* New York Heart Association (NYHA) cardiac function classification of grade II or III at screening
* Other Criteria apply, please contact the investigator

Exclusion Criteria:

* Patients with cardiac devices such as pacemakers, implantable cardioverter defibrillators (ICDs), or cardiac resuscitation-enabled implantable cardioverter defibrillators (CRT-Ds)
* Patients with heart failure due to the primary disease hypertrophic cardiomyopathy (including the dilated phase), restrictive cardiomyopathy, amyloidosis, takotsubo cardiomyopathy, congenital heart disease, cardiac sarcoidosis, or constrictive pericarditis
* Other Criteria apply, please contact the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 26 weeks post-transplant
  Adverse events and safety in the 26 weeks after HS-005 administration

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction in Cardiac MRI scan | 26 weeks and 52 weeks post-transplant
  Left Ventricular Ejection Fraction in the 26 weeks and 52 weeks after HS-005 administration
Left Ventricular Ejection Fraction in Echocardiography | 26 weeks and 52 weeks post-transplant
  Left Ventricular Ejection Fraction in the 26 weeks and 52 weeks after HS-005 administration
Left Ventricular volume in Cardiac MRI scan | 26 weeks and 52 weeks post-transplant
  Left Ventricular volume in the 26 weeks and 52 weeks after HS-005 administration
Left Ventricular volume in Echocardiography | 26 weeks and 52 weeks post-transplant
  Left Ventricular volume in the 26 weeks and 52 weeks after HS-005 administration
Myocardial wall motion evaluation in MRI | 26 weeks and 52 weeks post-transplant
  Myocardial wall motion evaluation (Index of myocardial strain) in the 26 weeks and 52 weeks
Myocardial wall motion evaluation in Echocardiography | 26 weeks and 52 weeks post-transplant
  Myocardial wall motion evaluation (Index of myocardial strain) in the 26 weeks and 52 weeks
Myocardial blood flow in SPECT | 26 weeks and 52 weeks post-transplant
  Myocardial blood flow in the 26 weeks and 52 weeks
Myocardial viability in SPECT | 26 weeks and 52 weeks post-transplant
  Myocardial viability in the 26 weeks and 52 weeks
6-minute walk distance | 26 weeks and 52 weeks post-transplant
  6-minute walk distance in the 26 weeks and 52 weeks
N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) | 26 weeks and 52 weeks post-transplant
  NT-proBNP measurement in the 26 weeks and 52 weeks
QoL questioner (Kansas City Cardiomyopathy Questionnaire) | 26 weeks and 52 weeks post-transplant
  KCCQ evaluation in the 26 weeks and 52 weeks
QoL questioner (EuroQol 5 dimensions 5-level) | 26 weeks and 52 weeks post-transplant
  EQ-5D-5L evaluation in the 26 weeks and 52 weeks

IPD SHARING:
Plan to Share IPD: No